CLINICAL TRIAL: NCT06054698
Title: A Multicenter, Randomized, Double-blind, Placebo-parallel-controlled, Phase II Clinical Study to Evaluate the Efficacy and Safety of HRS9531 Injection in Overweight or Obese Subjects
Brief Title: Efficacy and Safety of HRS9531 Injections in Overweight or Obese Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS9531-203
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS9531 injection (Experimental)
  Interventions: Drug: HRS9531 injection
- HRS9531 injection Placebo (Placebo Comparator)
  Interventions: Drug: HRS9531 injection Placebo

INTERVENTIONS:
Drug: HRS9531 injection — HRS9531 injection , QW，36 weeks
  Arms: HRS9531 injection
Drug: HRS9531 injection Placebo — HRS9531 injection Placebo，QW，36 weeks
  Arms: HRS9531 injection Placebo

SUMMARY:
To assess the efficacy of HRS9531 injection compared with placebo in weight reduction in overweight or obese subjects after 36 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. Male or female subjects, 18-65 years of age at the time of signing informed consent.
3. 28.0 ≤BMI≤ 40.0 kg/m2 or 24 ≤BMI< 28.0 kg/m2 with at least 1 weight-related comorbidity at screening visit.
4. Diet and exercise control for at least 3 months before screening visit, and less than 5 kg self-reported change within the last 3 months.

Exclusion Criteria:

1. Presence of - clinically significant lab or ECG results that may affect the evaluation of the efficacy or safety of the study drug at screening visit.
2. poor-controlled hypertension.
3. PHQ-9 score ≥15.
4. Medical history of illness that affects weight.
5. History of diabetes.
6. Acute infection, acute trauma, or medium to large surgery within 1 month prior to screening.
7. History of acute cardiovascular and cerebrovascular diseases.
8. Any organ-system malignancies developed within 5 years except cured local basal cell carcinoma of skin and cervical carcinoma in situ.
9. Confirmed or suspected depression, bipolar disorder, suicidal tendency, schizophrenia, or other serious mental illness.
10. History of alcohol , medication or drug abuse within 1 year prior to screening.
11. Use of any medication or treatment that may cause significant weight change within 3 months.
12. History of bariatric surgery.
13. Subjects participating in QT/QTc studies need to comply with relevant examinations.
14. Known or suspected hypersensitivity to trial product(s) or related products.
15. Participation in other clinical trials within 3 month prior to screening.
16. History of blood donation or blood loss in the 3 months before screening, or blood transfusion in the 2 months before screening
17. Surgery is planned during the trial.
18. Mentally incapacitated or speech-impaired.
19. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method.
20. Researchers and relevant staff of the research Centre or other people directly involved in the implementation of the programme, and their immediate family members.
21. In the judgment of the investigator, there are circumstances that affect the safety of the subject or any other interference with the evaluation of the test results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight | Week 0, Week 36

SECONDARY OUTCOMES:
Proportion of Subjects with weight loss of ≥5% from baseline in body weight after 36 weeks of treatment | Week 36
Proportion of Subjects with weight loss of ≥10% from baseline in body weight after 36 weeks of treatment | Week 36
Proportion of Subjects with weight loss of ≥15% from baseline in body weight after 36 weeks of treatment | Week 36
Change from baseline in body weight after 36 weeks of treatment | Week 0, Week 36
Change from baseline in waist circumference after 36 weeks of treatment | Week 0, Week 36
Change from baseline in BMI after 36 weeks of treatment | Week 0, Week 36
Change from baseline in blood pressure after 36 weeks of treatment | Week 0, Week 36
Change from baseline in total cholesterol after 36 weeks of treatment | Week 0, Week 36
Change from baseline in fasting plasma glucose (FPG) after 36 weeks of treatment | Week 0, Week36
Change from baseline in glycosylated haemoglobin (HbA1c) after 36 weeks of treatment | Week 0, Week 36
Number of AEs During the Trial | Week 0 to Week 36

IPD SHARING:
Plan to Share IPD: Undecided